CLINICAL TRIAL: NCT04623138
Title: A Decentralized, Prospective Study Exploring the Relationship Between Passively-collected Data From Wearable Activity Devices and SARS-CoV-2 Infection
Brief Title: A Virtual Prospective Study Exploring Activity Trackers and COVID-19 Infections
Status: Completed | Type: Observational
Sponsor: Evidation Health (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Eli Lilly and Company (Industry); Bill and Melinda Gates Foundation (Other); Vir Biotechnology, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: COVID Signals
Record Dates: First submitted 2020-10-30; First posted 2020-11-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: COVID-19; SARS-Cov Infection; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The Phosphorus COVID-19 RT-qPCR Test will be used for the qualitative detection of nucleic acid from SARS-CoV-2 in saliva specimens that are either self-collected at home or in a healthcare setting using the Oragene Dx OGD-510 collection device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Garmin Study Device Group: Individuals who are randomly assigned to receive the Garmin vívosmart® 4
- Empatica Study Device Group: Individuals who are randomly assigned to receive the Empatica E4

SUMMARY:
Prospective, observational, exploratory study exploring the relationship between passively-collected data from wearable activity devices and SARS-CoV-2 infection

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+ years of age
* Lives in the United States
* Speaks, reads, and understands English
* Willing and able to use and wear a wrist-worn activity device daily, during the day and during sleep, or as much as is possible, for the duration of the study
* Meets minimum software and device requirements for the wrist-worn activity device (Apple iOS 12 and up, Android version 6.0 and up)
* Willing to answer daily, weekly and monthly surveys for the duration of the study
* Willing to provide weekly self-collected saliva samples, plus one additional sample if prompted to do so (up to 9 total samples), and ship back the sample(s) within 24 hours of sample collection

Exclusion Criteria:

* Self-reported previous diagnosis of COVID-19
* Currently participating in any type of clinical trial
* Lives in the District of Columbia (Washington D.C.), Alaska, Hawaii, Arizona, Nevada, U.S. military base located overseas, or U.S. territories (Puerto Rico, U.S. Virgin Islands, Guam, Northern Mariana Island, or American Samoa)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants (ages 18+) who reside in the contiguous United States and are at elevated risk of contracting COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Development of database containing physiological, behavioral data in combination with SARS-CoV-2 infection | Through study completion, an average of 7 months
  To develop a database of physiological and behavioral data via wearable devices and self-reported questionnaires (e.g.,symptoms) combined with laboratory confirmation of SARS- CoV-2 infection.
Correlation between SARS-CoV-2 infection and collected wearable data and self-reported data | Through study completion, an average of 7 months
  Physiological and behavioral data from wearable devices (Garmin vivosmart 4, Empatica E4) , patient self-reported data questionnaires (includes but is not limited to demographics, symptoms, medical history, lifestyle, comorbidities, and Medical care utilization), and laboratory diagnostic confirmation of SARS-CoV-2 infection.

SECONDARY OUTCOMES:
Lift of the analytical models as expressed as the ratio of COVID-19+ recall (COVID-19+ cases detected by model as a percentage of total positive cases)/Healthy false positives (healthy cases detected by the model as being COVID-19+). | Through study completion, an average of 7 months
  Lift is a measure of model performance and will be evaluated at multiple timepoints along the infection time-course (for example, 1 day prior to illness onset, onset, day 3, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Ramirez, PhD, Principal Investigator — Evidation Health; Luca Foschini, PhD, Principal Investigator — Evidation Health
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Background] Arons MM, Hatfield KM, Reddy SC, Kimball A, James A, Jacobs JR, Taylor J, Spicer K, Bardossy AC, Oakley LP, Tanwar S, Dyal JW, Harney J, Chisty Z, Bell JM, Methner M, Paul P, Carlson CM, McLaughlin HP, Thornburg N, Tong S, Tamin A, Tao Y, Uehara A, Harcourt J, Clark S, Brostrom-Smith C, Page LC, Kay M, Lewis J, Montgomery P, Stone ND, Clark TA, Honein MA, Duchin JS, Jernigan JA; Public Health-Seattle and King County and CDC COVID-19 Investigation Team. Presymptomatic SARS-CoV-2 Infections and Transmission in a Skilled Nursing Facility. N Engl J Med. 2020 May 28;382(22):2081-2090. doi: 10.1056/NEJMoa2008457. Epub 2020 Apr 24. PMID 32329971
- [Background] Gandhi M, Yokoe DS, Havlir DV. Asymptomatic Transmission, the Achilles' Heel of Current Strategies to Control Covid-19. N Engl J Med. 2020 May 28;382(22):2158-2160. doi: 10.1056/NEJMe2009758. Epub 2020 Apr 24. No abstract available. PMID 32329972
- [Background] CDC COVID-19 Response Team. Preliminary Estimates of the Prevalence of Selected Underlying Health Conditions Among Patients with Coronavirus Disease 2019 - United States, February 12-March 28, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):382-386. doi: 10.15585/mmwr.mm6913e2. PMID 32240123
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Chow EJ, Schwartz NG, Tobolowsky FA, Zacks RLT, Huntington-Frazier M, Reddy SC, Rao AK. Symptom Screening at Illness Onset of Health Care Personnel With SARS-CoV-2 Infection in King County, Washington. JAMA. 2020 May 26;323(20):2087-2089. doi: 10.1001/jama.2020.6637. PMID 32301962
- [Background] Han C, Duan C, Zhang S, Spiegel B, Shi H, Wang W, Zhang L, Lin R, Liu J, Ding Z, Hou X. Digestive Symptoms in COVID-19 Patients With Mild Disease Severity: Clinical Presentation, Stool Viral RNA Testing, and Outcomes. Am J Gastroenterol. 2020 Jun;115(6):916-923. doi: 10.14309/ajg.0000000000000664. PMID 32301761
- [Background] Menni C, Valdes AM, Freidin MB, Sudre CH, Nguyen LH, Drew DA, Ganesh S, Varsavsky T, Cardoso MJ, El-Sayed Moustafa JS, Visconti A, Hysi P, Bowyer RCE, Mangino M, Falchi M, Wolf J, Ourselin S, Chan AT, Steves CJ, Spector TD. Real-time tracking of self-reported symptoms to predict potential COVID-19. Nat Med. 2020 Jul;26(7):1037-1040. doi: 10.1038/s41591-020-0916-2. Epub 2020 May 11. PMID 32393804
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Poyiadji N, Shahin G, Noujaim D, Stone M, Patel S, Griffith B. COVID-19-associated Acute Hemorrhagic Necrotizing Encephalopathy: Imaging Features. Radiology. 2020 Aug;296(2):E119-E120. doi: 10.1148/radiol.2020201187. Epub 2020 Mar 31. No abstract available. PMID 32228363
- [Background] Landa N, Mendieta-Eckert M, Fonda-Pascual P, Aguirre T. Chilblain-like lesions on feet and hands during the COVID-19 Pandemic. Int J Dermatol. 2020 Jun;59(6):739-743. doi: 10.1111/ijd.14937. Epub 2020 Apr 24. No abstract available. PMID 32329897
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Grady, D. (2020, June 11). Covid-19 Patient Gets Double Lung Transplant, Offering Hope for Others. Retrieved from https://www.nytimes.com/2020/06/11/health/coronavirus-lung-transplant.html
- [Background] Grant MC, Geoghegan L, Arbyn M, Mohammed Z, McGuinness L, Clarke EL, Wade RG. The prevalence of symptoms in 24,410 adults infected by the novel coronavirus (SARS-CoV-2; COVID-19): A systematic review and meta-analysis of 148 studies from 9 countries. PLoS One. 2020 Jun 23;15(6):e0234765. doi: 10.1371/journal.pone.0234765. eCollection 2020. PMID 32574165
- [Background] Shapiro A, Marinsek N, Clay I, Bradshaw B, Ramirez E, Min J, Trister A, Wang Y, Althoff T, Foschini L. Characterizing COVID-19 and Influenza Illnesses in the Real World via Person-Generated Health Data. Patterns (N Y). 2020 Dec 13;2(1):100188. doi: 10.1016/j.patter.2020.100188. eCollection 2021 Jan 8. PMID 33506230
- [Background] Auwaerter, PA. "Coronavirus COVID-19 (SARS-CoV-2)." Johns Hopkins ABX Guide, Johns Hopkins Medicine, 2020. https://www.hopkinsguides.com/hopkins/view/Johns_Hopkins_ABX_Guide/540 747/all/Coronavirus_COVID_19__SARS_CoV_2_#2
- See also: Statement on the second meeting of the International Health Regulations (2005) Emergency Committee regarding the outbreak of novel coronavirus (2019-nCoV). (n.d.) — http://www.who.int/news-room/detail/30-01-2020-statement-on-the-second-meeting-of-the-international-health-regulations-(2005)-emergency-committee-regarding-the-outbreak-of-novel-coronavirus-(2019-ncov)
- See also: COVID-19 Map. (n.d.) — https://coronavirus.jhu.edu/map.html
- See also: Modes of transmission of virus causing COVID-19: Implications for IPC precaution recommendations. (n.d.). — https://www.who.int/news-room/commentaries/detail/modes-of-transmission-of-virus-causing-covid-19-implications-for-ipc-precaution-recommendations
- See also: Coronavirus disease 2019 (COVID-19) Situation Report - 73 (Issue brief No. 73). — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200402-sitrep-73-covid-19.pdf?sfvrsn=5ae25bc7_6
- See also: World Health Organization. (2020, April 1). COVID-19 - Virtual Press Conference [Press release]. — https://www.who.int/docs/default-source/coronaviruse/transcripts/who-audio-emergencies-coronavirus-press-conference-full-01apr2020-final.pdf?sfvrsn=573dc140_2
- See also: UCSF TemPredict Study. (n.d.). — https://ouraring.com/ucsf-tempredict-study
- See also: COVID-19 Wearables Study. (n.d.). — https://innovations.stanford.edu/wearables
- See also: Coronavirus. (n.d.) — https://www.who.int/health-topics/coronavirus#tab=tab_3
- See also: Phosphorus COVID-19 RT-QPCR Test - Letter of Authorization — http://www.fda.gov/media/138652/download
- See also: Oragene-Dx OGD-510 — https://www.dnagenotek.com/US/pdf/PD-BR-00041.pdf
- See also: Coronavirus Disease 2019 (COVID-19) 2020 Interim Case Definition, Approved April 5, 2020 — http://ndc.services.cdc.gov/case-definitions/coronavirus-disease-2019-2020/